CLINICAL TRIAL: NCT01560637
Title: Open-Label Extension Study of UT-15C in Subjects With Pulmonary Arterial Hypertension- A Long-Term Follow-Up to Protocol TDE-PH-310
Brief Title: An Open-Label, Long-Term Study of Oral Treprostinil in Subjects With Pulmonary Arterial Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TDE-PH-311
Record Dates: First submitted 2012-03-09; First posted 2012-03-22 (Estimated); Results first posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: PAH; PH; FREEDOM; 6 minute walk test; treprostinil; open label
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — treprostinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- UT-15C (Experimental): Open label access
  Interventions: Drug: UT-15C (treprostinil diolamine)

INTERVENTIONS:
Drug: UT-15C (treprostinil diolamine) — UT-15C extended release oral tablet three times daily

SUMMARY:
This study is an international, multi-center, open-label study designed to provide oral treprostinil (UT-15C) to eligible subjects with pulmonary arterial hypertension who have completed the TDE-PH-310 study. The purpose of this study is to assess the long-term safety of UT-15C and to assess the effects of long-term treatment with UT-15C on exercise capacity.

ELIGIBILITY:
Inclusion Criteria:

* Participated in United Therapeutics Study TDE-PH-310
* All women of childbearing potential (WOCBP) must have practiced true abstinence from intercourse when it was in line with their preferred and usual lifestyle or used 2 different forms of highly effective contraception for the duration of the study and for at least 30 days after discontinuing study medication.
* Males who participated in the study must have used a condom during the length of the study and for at least 48 hours after their last dose of study medication.

Exclusion Criteria:

* The subject was pregnant or lactating.
* The subject had received infused or inhaled prostacyclin therapy for 29 days or more.
* The subject was prematurely discontinued from TDE-PH-310 for reasons other than a clinical worsening event.
* The subject developed a concurrent illness or condition during the conduct of TDE-PH-310 which, in the opinion of the Investigator, would represent a risk to their overall health if they enrolled in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 471 (Actual)
Dates: Start 2013-09-11 (Actual); Primary Completion 2021-08-12 (Actual); Study Completion 2021-08-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (153):
- United States (38):
  - Arizona Pulmonary Specialists, Ltd., Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - University of California, San Francisco-Fresno, Fresno, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California-Davis Medical Group, Advanced Lung Disease/Transplant Program, Sacramento, California
  - David Geffen School of Medicine, Torrance, California
  - University of Colorado Hospital, Aurora, Colorado
  - University of Florida, Gainesville, Florida
  - University of Florida College of Medicine Jacksonville- Division of Pulmonary & Critical Medicine, Jacksonville, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - Piedmont - Georgia Lung Associates, Austell, Georgia
  - HeartCare Midwest, Peoria, Illinois
  - Indiana University Hospital, Carmel, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Kentuckiana Pulmonary Associates, Louisville, Kentucky
  - University of Maryland, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Beaumont Health, Troy, Michigan
  - Nebraska Medical Center, Omaha, Nebraska
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - University of Rochester, Rochester, New York
  - Asheville Cardiology Associates, Asheville, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - University Hospital, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Legacy Research Institute, Portland, Oregon
  - Perelman Center for Advanced Medicine, University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center - Presbyterian Cardiovascular Institute, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Sentara Cardiovascular Research Institute, Norfolk, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
- Argentina (5):
  - Sanatorio San José, CABA, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires, Distrito Federal
  - Hospital Italiano Garibaldi, Rosario, Santa Fe Province
  - Sanatorio de la Trinidad Mitre, Buenos Aires
  - Hospital Dr. José María Cullen, Santa Fe
- Australia (8):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - Saint Vincents Hospital, Sydney, New South Wales
  - Macquarie University, Sydney, New South Wales
  - Prince Charles Hospital, Chermside, Queensland
  - Royal Hobart Hospital, Hobart, Tasmania
  - The Alfred Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- Austria (2):
  - Krankenhaus Elisabethinen Linz, Linz, Upper Austria
  - Medizinische Universität Wien, Vienna
- Brazil (8):
  - Hospital das Clinicas da Universidade Federal de Goias, Goiânia, Goiás
  - Hospital das Clínicas da Universidade Federal de Minas Gerais, Belo Horizonte, Minas Gerais
  - Hospital Madre Teresa, Belo Horizonte, Minas Gerais
  - Complexo Hospitalar Santa Casa de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital das Clínicas da Faculdade de Medicina de Botucatu- UNESP, Botucatu, São Paulo
  - Hospital da Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo
  - Escola Paulista de Medicina, Universidade Federal de São Paulo, São Paulo, São Paulo
  - Hospital Alemão Oswaldo Cruz, São Paulo
- Canada (4):
  - Respiratory Research Foundation, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Vancouver Coastal Health, Vancouver, British Columbia
  - Lawson Health Research Institute, London, Ontario
- Chile (2):
  - Centro de Investigaciones TASOL, Santiago, Santiago Metropolitan
  - Clínica Tabancura, Vitacura, Santiago Metropolitan
- China (16):
  - Beijing Chao-Yang Hospital, Beijing, Beijing Municipality
  - Guangdong General Hospital, Guangzhou, Guangdong
  - Wuhan Asia Heart Hospital, Wuhan, Hubei
  - Xiangya Hospital, Changsha, Hunan
  - The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanchang Medical University, Nanchang, Jiangxi
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Renji Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - West China Hospital, Chengdu, Sichuan
  - Peking Union Medical College Hospital, Beijing
  - Beijing Shijitan Hospital, Beijing
  - Chinese PLA General Hospital, Beijing
  - The Affiliated Hospital of Qingdao University, Qingdao
  - Renji Hospital of Shanghai Jiaotong University, Shanghai
  - Shanghai Pulmonary Hospital of Tongji University, Shanghai
  - Shenyang General Hospital of Shenyang Military Command, Shenyang
- Denmark (2):
  - Aarhus Universitetshospital, Skejby, Aarhus
  - Rigshospitalet-Copenhagen University Hospital, Copenhagen
- France (6):
  - Hopital Haut-Leveque, CHU Bordeaux, Pessac, Aquitaine
  - Hopital Jean Minjoz Centre Hospitalier Universitaire Besancon, Besançon, Franche-comte
  - Centre Hospitalier Régional Universitaire de Lille - Hôpital Claude Huriez, Lille, Hauts-de-France
  - CHU de Montpellier, Montpellier, Languedoc-roussillon
  - Hopital Brabois, Vandœuvre-lès-Nancy, Limousin, Lorraine
  - Centre Hospitalier Universitaire Hopital Nord, Marseille, Provence-Alpes-Côte d'Azur Region
- Germany (13):
  - Thoraxklinik am Universitätsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Ludwig-Maximilians-Universitat Munchen, München, Bavaria
  - Universitätsklinikum Regensburg, Regensburg, Bavaria
  - Missionsarztliche Klinik Wurzburg gGmbH, Würzburg, Bavaria
  - Universitätsmedizin Greifswald, Greifswald, Mecklenburg-Vorpommern
  - Bergmannsheil Berufsgenossenschaftliche Universitätsklinik GmbH, Bochum, North Rhine-Westphalia
  - Universitätsklinikum Köln, Cologne, North Rhine-Westphalia
  - Herzzentrum Duisburg, Duisburg, North Rhine-Westphalia
  - Universitätsmedizin der Johannes Gutenberg Universität, Mainz, Rhineland-Palatinate
  - Universitätsklinikum des Saarlandes, Homburg, Saarland
  - Technische Universität Dresden, Dresden, Saxony
  - Universitätsklinikum Leipzig, Leipzig, Saxony
  - Universitätskrankenhaus Hamburg-Eppendorf, Hamburg
- Greece (2):
  - University General Hospital of Attikon, Athens, Attica
  - General Hospital of Thessaloniki, "G.Papanikolaou", Thessaloniki, Macedoni
- India (13):
  - CARE Hospital, Hyderabad, Andhra Pradesh
  - Mediciti Hospital, Hyderabad, Andhra Pradesh
  - Care Institute Medical Sciences, Ahmedabad, Gujarat
  - Apollo Hospitals International, Ltd., Gandhinagar, Gujarat
  - Medanta - The Medicity, Gurgaon, Haryana
  - Narayana Institute of Cardiac Sciences, Bangalore, Karnataka
  - KEM Hospital, Mumbai, Maharashtra
  - King Edward Memorial Hospital & Seth Gordhandas Sunderdas Medical College, Mumbai, Maharashtra
  - Ruby Hall Clinic, Pune, Maharashtra
  - Sir Ganga Ram Hospital, New Delhi, National Capital Territory of Delhi
  - Indraprastha Apollo Hospital, New Delhi, National Capital Territory of Delhi
  - Apollo Hospital, Chennai, Tamil Nadu
  - G. Kuppuswamy Naidu Memorial Hospital, Coimbatore, Tamil Nadu
- Israel (5):
  - Rabin Medical Center, Petach Tikvah, Petah Tiqwa
  - The Chaim Sheba Medical Center at Tel Hashomer, Tel Litwinsky, Tel Aviv
  - Rambam Health Corp., Haifa
  - Carmel Medical Center, Haifa
  - Hadassah Medical Center, Jerusalem
- Italy (4):
  - Azienda Ospedaliera Universitaria, Napoli
  - Istituto Mediterraneo Trapianti e Terapia Alta Specializzazione (ISMETT), Palermo
  - Fondazione IRCCS Policlinico S. Matteo, Pavia
  - Azienda Policlinico Umberto I di Roma, Roma
- Mexico (2):
  - Instituto Nacional de Cardiologia Ignacio Chavez, Tlalpan, Mexico City
  - Unidad de Investigacion Clinica en Medicina S.C., Monterrey, Nuevo León
- Netherlands (2):
  - Universitair Medisch Centrum Sint Radboud, Nijmegen, Gelderland
  - Vrije Universiteit Medisch Centrum, Amsterdam, North Holland
- Poland (4):
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok
  - Szpital Kliniczny Przemienienia Panskiego Uniwersytetu Medycznego im K. Marcinkowskiego w Poznaniu, Krakow
  - Krakowski Szpital Specjalistyczny im. Jana Pawla II, Małogoskie
  - Europejskie Centrum Zdrowia Otwock, Szpital im. Fryderyka Chopina, Otwock
- Singapore (2):
  - National University Hospital, Singapore
  - National Heart Centre Singapore, Singapore
- South Korea (5):
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg, Västra Götaland County
  - Karolinska University Hospital Solna, Stockholm
- Taiwan (4):
  - National Cheng Kung University Hospital, Tainan, Tainan CITY
  - Veterans General Hospital-Kaohsiung, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
- United Kingdom (4):
  - Papworth Hospital, Papworth Everard, Cambridgshire
  - Royal Free Hospital, London, England
  - Freeman Hospital, Newcastle upon Tyne, England
  - Royal Hallamshire Hospital, Sheffield, England

REFERENCES:
- [Derived] Grunig E, Rahaghi F, Elwing J, Vizza CD, Pepke-Zaba J, Shen J, Yao H, Hage A, Rosenkranz S, Vonk M, Balasubramanian V, Yuanhua Y, Yu Z, Lordan J, Cadaret L, Grover R, Ousmanou A, Seaman S, Deng C, Broderick M, White RJ; FREEDOM-EV Investigators. Oral Treprostinil is Associated with Improved Survival in FREEDOM-EV and its Open-Label Extension. Adv Ther. 2024 Feb;41(2):618-637. doi: 10.1007/s12325-023-02711-x. Epub 2023 Dec 6. PMID 38055186

RESULTS

PARTICIPANT FLOW:
Groups:
- UT-15C: Open label access
  UT-15C (treprostinil diethanolamine): UT-15C sustained release oral tablet for three times daily administration
Period: Overall Study
Arm/Group | UT-15C
Started | 470 (471 subjects from the parent study (TDE-PH-310) consented to participate in TDE-PH-311. However, one subject withdrew consent prior to receiving oral treprostinil in TDE-PH-311. This subject was not included in the data summary.)
Completed | 272
Not Completed | 198
Not completed — Adverse Event | 63
Not completed — Death | 69
Not completed — Lost to Follow-up | 8
Not completed — Protocol Violation | 8
Not completed — Withdrawal by Subject | 24
Not completed — Progressive Disease | 20
Not completed — Other Reason Not Specified | 6

BASELINE CHARACTERISTICS:
Population: All 470 subjects who received oral treprostinil during this study are included in the Baseline Analysis Population.
Arm/Group | UT-15C
Number analyzed (Participants) | 470
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 398
  >=65 years | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.2 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 374
  Male | 96
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 135
  Not Hispanic or Latino | 334
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 213
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 245
  More than one race | 0
  Unknown or Not Reported | 2
Etiology of Pulmonary Arterial Hypertension (PAH) [Count of Participants; unit: Participants]
  Idiopathic of Heritable PAH | 299
  Collagen Vascular Disease | 114
  HIV Infection | 8
  Congenital Heart Defect | 38
  Other | 11
Background PAH Therapy at Randomization in Parent Study [Count of Participants; unit: Participants]
  Phosphodiesterase Type 5 Inhibitor (PDE5-I) Alone/Soluble Guanylate Cyclase (sGC) Stimulator Alone | 348
  Endothelin Receptor Antagonist (ERA) alone | 122
Time since Diagnosis [Mean (Standard Deviation); unit: years] | 3.16 (2.69)
6-Minute Walk Distance (6MWD) at Baseline [Mean (Standard Deviation); unit: meters] | 392.0 (128.1)
WHO Functional Class at Baseline [Count of Participants; unit: Participants] — The World Health Organization functional classification (WHO-FC) is a clinician-rated assessment used widely to assess PAH severity and functioning.
  Class I (least severe): Patients are without limitation of physical activity.
  Class II: Patients are comfortable at rest. Ordinary physical activity causes undue dyspnea or fatigue, chest pain or near syncope.
  Class III: Marked limitation of physical activity. They are comfortable at rest.
  Class IV (most severe): Inability to carry out any physical activity without symptoms. These patients manifest signs of right heart failure.
  Participants
    I | 41
    II | 226
    III | 182
    IV | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events
Description: All subjects who received oral treprostinil in TDE-PH-311 were included in the Safety population. All AEs were captured from the time the ICF was signed. All AEs were followed until resolution (or return to normal or baseline values), until they were judged by the Investigator to no longer be clinically significant, or for up to 30 days if the AE extended beyond the final visit. All SAEs were followed until resolution, death, or the subject was lost to follow-up, even if they were ongoing more than 30 days after completion of the final visit. The overall summary of AEs includes the number of subjects with any AE, the number of subjects with any study drug-related AEs, the number of subjects with AEs leading to study drug withdrawal, the number of subjects with any serious AEs, the number of subjects with any severe AEs, and the number of subjects with any study drug-related severe/serious AEs. AEs were coded using the Medical Dictionary for Regulatory Activities.
Time Frame: Participants will be followed every 12 weeks, at minimum, until they discontinue the study or the study is discontinued by the sponsor or for a period up to 2.5 years
Population: All subjects who received oral treprostinil in TDE-PH-311 were included in the Safety population.
Measure: Number; unit: events
Arm/Group | UT-15C
Number analyzed (Participants) | 470
events
  Adverse Event | 450
  Study Drug Related AE | 362
  AE Leading to Study Drug Withdrawal | 126
  Serious AE | 206
  Severe AE | 182
  Study Drug Related Severe AE | 67
  Study Drug Related Serious AE | 37

2. Secondary Outcome: Change in 6-Minute Walk Distance From Baseline
Description: A summary of change from Baseline in 6MWD at Week 48 for the Safety Population is provided. The Safety Population is all subjects who received oral treprostinil in TDE-PH-311.
Time Frame: Baseline to Week 48
Population: All participants are subjects who received oral treprostinil in TDE-PH-311. For post-Baseline visits, only subjects with measurements at Baseline and the corresponding visit are included. Baseline is defined as the last measurement prior to the first dose of oral treprostinil in TDE-PH-311.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | UT-15C
Number analyzed (Participants) | 341
meters | 20.1 (79.6)

3. Secondary Outcome: Change in Borg Dyspnea Score From Baseline to Week 48
Description: Change in Borg Dyspnea Score from at Week 48 is provided for the Safety Population (all subjects who received oral treprostinil in TDE-PH-311).
  The Borg Dyspnea Scale is a 0 to 10 rated numerical score used to measure dyspnea as reported by the patient during submaximal exercise and was administered during six-minute walk testing (6MWT), one of the most common and frequently used measures to assess disease severity in PAH. The numbers on the scale are as follows: 0 (no shortness of breath [SOB]), 0.5 (very very slight SOB), 1 (very slight SOB), 3 (moderate SOB), 4 (somewhat severe SOB), 5 (severe SOB), 7 (very severe SOB), 9 (very very severe SOB), 10 (maximal SOB).
Time Frame: Baseline to Week 48
Population: Safety Population (all subjects who received oral treprostinil in TDE-PH-311). For post-Baseline visits, only subjects with measurements at Baseline and the corresponding visit are included. Baseline is defined as the last measurement prior to the first dose of oral treprostinil in TDE-PH-311.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | UT-15C
Number analyzed (Participants) | 341
score on a scale | -0.49 (1.92)

4. Secondary Outcome: Change From Baseline to Week 48 in WHO Functional Class
Description: Change from Baseline at Week 48 in WHO FC in the Safety Population (all subjects who received oral treprostinil in TDE-PH-311).
  The World Health Organization functional classification (WHO-FC) is a clinician-rated assessment used widely to assess PAH severity and functioning.
  Class I (least severe): Patients are without limitation of physical activity.
  Class II: Patients are comfortable at rest. Ordinary physical activity causes undue dyspnea or fatigue, chest pain or near syncope.
  Class III: Marked limitation of physical activity. They are comfortable at rest.
  Class IV (most severe): Inability to carry out any physical activity without symptoms. These patients manifest signs of right heart failure.
Time Frame: Baseline to Week 48
Population: Safety Population was analyzed. Baseline is defined as the last measurement prior to the first dose of oral treprostinil in TDE PH 311.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | UT-15C
Number analyzed (Participants) | 362
score on a scale | -0.2 (0.6)

5. Secondary Outcome: Change in N-terminal Pro-brain Natriuretic Peptide (NT-proBNP) From Baseline to Week 48
Description: Change in N-terminal pro-brain natriuretic peptide from Baseline at Week 48 for the Safety Population (any subject who received oral treprostinil in TDE-PH-311)
Time Frame: Baseline to Week 48
Population: Subjects in the Safety Population were analyzed. For post-Baseline visits, only subjects with measurements at Baseline and the corresponding visit are included. Baseline is defined as the last measurement prior to the first dose of oral treprostinil in TDE-PH-311.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | UT-15C
Number analyzed (Participants) | 322
pg/mL | -179.23 (1968.99)

ADVERSE EVENTS:
Time Frame: AEs were recorded for each subject throughout the course of the study from Baseline to 30 days following the final study visit (up to 356 weeks).
Description: All AEs were captured from the time the ICF was signed. All AEs were followed until resolution (or return to baseline values), until they were judged by the Investigator to no longer be clinically significant, or for up to 30 days if the AE extended beyond the final visit. All SAEs were followed until resolution, death, or the subject was lost to follow-up, even if they were ongoing more than 30 days after completion of the final visit.
Arm/Group | UT-15C
All-Cause Mortality (participants affected / at risk) | 74/470
Serious Adverse Events (participants affected / at risk) | 206/470
Other Adverse Events (participants affected / at risk) | 467/470
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | UT-15C (N=470)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 57 (79)
Pneumonia (Infections and infestations) | 32 (39)
Right ventricular failure (Cardiac disorders) | 22 (27)
Cardiac failure (Cardiac disorders) | 19 (25)
Septic shock (Infections and infestations) | 9 (9)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Acute kidney injury (Renal and urinary disorders) | 7 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Diarrhoea (Gastrointestinal disorders) | 6 (6)
Gastroenteritis (Infections and infestations) | 6 (6)
Hypotension (Vascular disorders) | 6 (6)
Anaemia (Blood and lymphatic system disorders) | 5 (5)
Cholecystitis acute (Hepatobiliary disorders) | 5 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Respiratory tract infection (Infections and infestations) | 5 (5)
Sepsis (Infections and infestations) | 5 (5)
Urinary tract infection (Infections and infestations) | 5 (5)
Cardiac arrest (Cardiac disorders) | 4 (4)
Cardiogenic shock (Cardiac disorders) | 4 (4)
Hyperthyroidism (Endocrine disorders) | 4 (4)
Syncope (Nervous system disorders) | 4 (4)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Appendicitis (Infections and infestations) | 3 (5)
Atrial fibrillation (Cardiac disorders) | 3 (3)
Atrial flutter (Cardiac disorders) | 3 (3)
COVID-19 (Infections and infestations) | 3 (3)
COVID-19 pneumonia (Infections and infestations) | 3 (3)
Cardiac failure congestive (Cardiac disorders) | 3 (3)
Cor pulmonale (Cardiac disorders) | 3 (3)
Fluid overload (Metabolism and nutrition disorders) | 3 (5)
Multiple organ dysfunction syndrome (General disorders) | 3 (3)
Myocardial infarction (Cardiac disorders) | 3 (3)
Shock (Vascular disorders) | 3 (3)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 3 (3)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (5)
Vomiting (Gastrointestinal disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Abortion induced (Surgical and medical procedures) | 2 (2)
Atrioventricular block complete (Cardiac disorders) | 2 (2)
Bronchitis (Infections and infestations) | 2 (2)
Cardiac failure acute (Cardiac disorders) | 2 (2)
Cardiopulmonary failure (Cardiac disorders) | 2 (2)
Catheterisation cardiac (Investigations) | 2 (2)
Cellulitis (Infections and infestations) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 2 (2)
Chest pain (General disorders) | 2 (3)
Clostridium difficile colitis (Infections and infestations) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Electrolyte imbalance (Metabolism and nutrition disorders) | 2 (3)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hand fracture (Injury, poisoning and procedural complications) | 2 (2)
Hepatic function abnormal (Hepatobiliary disorders) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2)
Melaena (Gastrointestinal disorders) | 2 (2)
Oedema (General disorders) | 2 (2)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Pericardial effusion (Cardiac disorders) | 2 (2)
Peritonitis (Infections and infestations) | 2 (2)
Pulmonary oedema (Cardiac disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Renal failure (Renal and urinary disorders) | 2 (2)
Right ventricular dysfunction (Cardiac disorders) | 2 (2)
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 2 (2)
Sudden death (General disorders) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1)
Acute abdomen (Gastrointestinal disorders) | 1 (1)
Acute hepatic failure (Hepatobiliary disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Acute pulmonary oedema (Cardiac disorders) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute right ventricular failure (Cardiac disorders) | 1 (1)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Adrenocortical insufficiency acute (Endocrine disorders) | 1 (1)
Amaurosis (Eye disorders) | 1 (1)
Anaemia of malignant disease (Blood and lymphatic system disorders) | 1 (1)
Aortic valve incompetence (Cardiac disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1)
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Atrioventricular block (Cardiac disorders) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1)
Bacterial translocation (Infections and infestations) | 1 (1)
Biliary tract disorder (Hepatobiliary disorders) | 1 (2)
Blood creatinine increased (Investigations) | 1 (1)
Brain injury (Nervous system disorders) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast mass (Reproductive system and breast disorders) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 1 (2)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Chest discomfort (General disorders) | 1 (1)
Cholecystitis infective (Infections and infestations) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Coagulation time prolonged (Investigations) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Coma (Nervous system disorders) | 1 (1)
Congestive hepatopathy (Hepatobiliary disorders) | 1 (1)
Cor pulmonale acute (Cardiac disorders) | 1 (2)
Coronary artery disease (Cardiac disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Diarrhoea infectious (Infections and infestations) | 1 (1)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Disease progression (General disorders) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (2)
Diverticulum (Gastrointestinal disorders) | 1 (1)
Endocrine ophthalmopathy (Eye disorders) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1)
Enteritis infectious (Infections and infestations) | 1 (1)
Erythropenia (Blood and lymphatic system disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (2)
Fibrocystic breast disease (Reproductive system and breast disorders) | 1 (1)
Gangrene (Infections and infestations) | 1 (1)
Gastric polyps (Gastrointestinal disorders) | 1 (1)
Gastric varices haemorrhage (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 1 (1)
Gastrointestinal vascular malformation haemorrhagic (Gastrointestinal disorders) | 1 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Generalised oedema (General disorders) | 1 (1)
Glomerulonephritis acute (Renal and urinary disorders) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hepatic cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1)
Hepatic encephalopathy (Hepatobiliary disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Infective exacerbation of bronchiectasis (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1)
Intermenstrual bleeding (Reproductive system and breast disorders) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 1 (2)
Liver injury (Hepatobiliary disorders) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lupus nephritis (Renal and urinary disorders) | 1 (1)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Mechanical ileus (Gastrointestinal disorders) | 1 (1)
Meningitis listeria (Infections and infestations) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1)
Metabolic encephalopathy (Metabolism and nutrition disorders) | 1 (1)
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Ophthalmic herpes zoster (Infections and infestations) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1)
POEMS syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Pelvic fluid collection (Reproductive system and breast disorders) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1)
Pneumonia aspiration (Infections and infestations) | 1 (1)
Pneumonia influenzal (Infections and infestations) | 1 (1)
Portal hypertensive gastropathy (Gastrointestinal disorders) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulseless electrical activity (Cardiac disorders) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Renal vasculitis (Renal and urinary disorders) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Scleroderma renal crisis (Renal and urinary disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Sialoadenitis (Infections and infestations) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Splenic rupture (Injury, poisoning and procedural complications) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 1 (1)
Subcapsular hepatic haematoma (Hepatobiliary disorders) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Sudden cardiac death (Cardiac disorders) | 1 (1)
Transaminases increased (Investigations) | 1 (1)
Tricuspid valve incompetence (Cardiac disorders) | 1 (1)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1)
Urinary bladder polyp (Renal and urinary disorders) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | UT-15C (N=470)
Anaemia (Blood and lymphatic system disorders) | 51 (55)
Thrombocytopenia (Blood and lymphatic system disorders) | 17 (19)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 9 (11)
Leukopenia (Blood and lymphatic system disorders) | 8 (10)
Splenomegaly (Blood and lymphatic system disorders) | 4 (4)
Coagulopathy (Blood and lymphatic system disorders) | 2 (2)
Pancytopenia (Blood and lymphatic system disorders) | 2 (2)
Anaemia of malignant disease (Blood and lymphatic system disorders) | 1 (1)
Antiphospholipid syndrome (Blood and lymphatic system disorders) | 1 (1)
Erythropenia (Blood and lymphatic system disorders) | 1 (1)
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1)
Hyperglobulinaemia (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Microcytic anaemia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (2)
Neutrophilia (Blood and lymphatic system disorders) | 1 (1)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 (1)
Splenic calcification (Blood and lymphatic system disorders) | 1 (1)
Splenic cyst (Blood and lymphatic system disorders) | 1 (1)
White blood cell disorder (Blood and lymphatic system disorders) | 1 (1)
Palpitations (Cardiac disorders) | 74 (81)
Right ventricular failure (Cardiac disorders) | 39 (54)
Cardiac failure (Cardiac disorders) | 26 (34)
Tachycardia (Cardiac disorders) | 11 (16)
Atrial fibrillation (Cardiac disorders) | 10 (11)
Atrial flutter (Cardiac disorders) | 7 (7)
Supraventricular tachycardia (Cardiac disorders) | 5 (5)
Cardiac arrest (Cardiac disorders) | 4 (4)
Cardiogenic shock (Cardiac disorders) | 4 (4)
Cor pulmonale (Cardiac disorders) | 4 (4)
Pericardial effusion (Cardiac disorders) | 4 (4)
Angina pectoris (Cardiac disorders) | 3 (3)
Cardiac failure congestive (Cardiac disorders) | 3 (4)
Extrasystoles (Cardiac disorders) | 3 (3)
Myocardial infarction (Cardiac disorders) | 3 (3)
Right ventricular dysfunction (Cardiac disorders) | 3 (4)
Supraventricular extrasystoles (Cardiac disorders) | 3 (3)
Aortic valve incompetence (Cardiac disorders) | 2 (2)
Arteriosclerosis coronary artery (Cardiac disorders) | 2 (2)
Atrioventricular block (Cardiac disorders) | 2 (2)
Atrioventricular block complete (Cardiac disorders) | 2 (2)
Atrioventricular block second degree (Cardiac disorders) | 2 (2)
Bradycardia (Cardiac disorders) | 2 (2)
Bundle branch block right (Cardiac disorders) | 2 (2)
Cardiac failure acute (Cardiac disorders) | 2 (2)
Cardiopulmonary failure (Cardiac disorders) | 2 (2)
Coronary artery disease (Cardiac disorders) | 2 (2)
Right ventricular hypertrophy (Cardiac disorders) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Acute right ventricular failure (Cardiac disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 1 (1)
Cardiac discomfort (Cardiac disorders) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 1 (3)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Cardiomegaly (Cardiac disorders) | 1 (1)
Cor pulmonale acute (Cardiac disorders) | 1 (2)
Pericarditis (Cardiac disorders) | 1 (1)
Pulseless electrical activity (Cardiac disorders) | 1 (1)
Sinus arrhythmia (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 1 (1)
Tricuspid valve incompetence (Cardiac disorders) | 1 (1)
Tricuspid valve stenosis (Cardiac disorders) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Atrial septal defect (Congenital, familial and genetic disorders) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 9 (9)
Vertigo (Ear and labyrinth disorders) | 9 (9)
Deafness (Ear and labyrinth disorders) | 5 (5)
Ear congestion (Ear and labyrinth disorders) | 2 (2)
Ear haemorrhage (Ear and labyrinth disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 1 (1)
Meniere's disease (Ear and labyrinth disorders) | 1 (1)
Middle ear inflammation (Ear and labyrinth disorders) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 18 (18)
Hyperthyroidism (Endocrine disorders) | 13 (15)
Adrenocortical insufficiency acute (Endocrine disorders) | 1 (1)
Cushingoid (Endocrine disorders) | 1 (1)
Eyelid oedema (Eye disorders) | 7 (7)
Conjunctival hyperaemia (Eye disorders) | 4 (4)
Vision blurred (Eye disorders) | 4 (4)
Visual impairment (Eye disorders) | 4 (4)
Cataract (Eye disorders) | 3 (4)
Amaurosis (Eye disorders) | 2 (2)
Dry eye (Eye disorders) | 2 (2)
Eye pruritus (Eye disorders) | 2 (2)
Blepharitis (Eye disorders) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 1 (1)
Conjunctivitis allergic (Eye disorders) | 1 (1)
Corneal bleeding (Eye disorders) | 1 (1)
Corneal erosion (Eye disorders) | 1 (1)
Diplopia (Eye disorders) | 1 (1)
Endocrine ophthalmopathy (Eye disorders) | 1 (1)
Exophthalmos (Eye disorders) | 1 (1)
Eye discharge (Eye disorders) | 1 (1)
Eye haemorrhage (Eye disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Keratitis (Eye disorders) | 1 (1)
Lacrimation increased (Eye disorders) | 1 (1)
Macular degeneration (Eye disorders) | 1 (1)
Ocular hyperaemia (Eye disorders) | 1 (1)
Periorbital oedema (Eye disorders) | 1 (1)
Periorbital pain (Eye disorders) | 1 (1)
Photophobia (Eye disorders) | 1 (1)
Pterygium (Eye disorders) | 1 (1)
Retinal haemorrhage (Eye disorders) | 1 (1)
Scleritis (Eye disorders) | 1 (1)
Ulcerative keratitis (Eye disorders) | 1 (1)
Vitreous floaters (Eye disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 311 (354)
Nausea (Gastrointestinal disorders) | 188 (197)
Vomiting (Gastrointestinal disorders) | 147 (161)
Abdominal pain (Gastrointestinal disorders) | 40 (43)
Abdominal pain upper (Gastrointestinal disorders) | 38 (40)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 36 (37)
Abdominal distension (Gastrointestinal disorders) | 35 (38)
Abdominal discomfort (Gastrointestinal disorders) | 30 (30)
Dyspepsia (Gastrointestinal disorders) | 28 (30)
Colitis (Gastrointestinal disorders) | 25 (29)
Constipation (Gastrointestinal disorders) | 22 (23)
Gastritis (Gastrointestinal disorders) | 22 (23)
Ascites (Gastrointestinal disorders) | 14 (14)
Dry mouth (Gastrointestinal disorders) | 10 (10)
Haemorrhoids (Gastrointestinal disorders) | 10 (10)
Irritable bowel syndrome (Gastrointestinal disorders) | 9 (9)
Toothache (Gastrointestinal disorders) | 9 (10)
Frequent bowel movements (Gastrointestinal disorders) | 8 (8)
Dysphagia (Gastrointestinal disorders) | 7 (7)
Diverticulum (Gastrointestinal disorders) | 6 (6)
Flatulence (Gastrointestinal disorders) | 5 (5)
Haematemesis (Gastrointestinal disorders) | 5 (5)
Melaena (Gastrointestinal disorders) | 5 (5)
Abdominal pain lower (Gastrointestinal disorders) | 4 (4)
Gingival bleeding (Gastrointestinal disorders) | 4 (4)
Haematochezia (Gastrointestinal disorders) | 4 (4)
Hiatus hernia (Gastrointestinal disorders) | 4 (4)
Oesophagitis (Gastrointestinal disorders) | 4 (4)
Chronic gastritis (Gastrointestinal disorders) | 3 (3)
Epigastric discomfort (Gastrointestinal disorders) | 3 (3)
Gastric polyps (Gastrointestinal disorders) | 3 (3)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3)
Large intestine polyp (Gastrointestinal disorders) | 3 (4)
Mouth ulceration (Gastrointestinal disorders) | 3 (3)
Portal hypertensive gastropathy (Gastrointestinal disorders) | 3 (3)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (5)
Anal incontinence (Gastrointestinal disorders) | 2 (2)
Dental caries (Gastrointestinal disorders) | 2 (2)
Enteritis (Gastrointestinal disorders) | 2 (2)
Faeces soft (Gastrointestinal disorders) | 2 (2)
Food poisoning (Gastrointestinal disorders) | 2 (2)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 2 (2)
Ileus (Gastrointestinal disorders) | 2 (2)
Inguinal hernia (Gastrointestinal disorders) | 2 (2)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (2)
Acute abdomen (Gastrointestinal disorders) | 1 (1)
Appendicitis noninfective (Gastrointestinal disorders) | 1 (1)
Defaecation urgency (Gastrointestinal disorders) | 1 (1)
Eructation (Gastrointestinal disorders) | 1 (1)
Gastric antral vascular ectasia (Gastrointestinal disorders) | 1 (1)
Gastric disorder (Gastrointestinal disorders) | 1 (1)
Gastric mucosal lesion (Gastrointestinal disorders) | 1 (1)
Gastric varices haemorrhage (Gastrointestinal disorders) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 1 (1)
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (2)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 (1)
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 1 (1)
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 1 (1)
Gastrointestinal vascular malformation haemorrhagic (Gastrointestinal disorders) | 1 (2)
Gingival swelling (Gastrointestinal disorders) | 1 (1)
Glossodynia (Gastrointestinal disorders) | 1 (1)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Mechanical ileus (Gastrointestinal disorders) | 1 (1)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1)
Pancreatic cyst (Gastrointestinal disorders) | 1 (1)
Peptic ulcer (Gastrointestinal disorders) | 1 (1)
Periodontal disease (Gastrointestinal disorders) | 1 (1)
Reflux gastritis (Gastrointestinal disorders) | 1 (1)
Retching (Gastrointestinal disorders) | 1 (1)
Salivary hypersecretion (Gastrointestinal disorders) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1)
Oedema peripheral (General disorders) | 85 (98)
Fatigue (General disorders) | 64 (68)
Chest pain (General disorders) | 45 (54)
Chest discomfort (General disorders) | 44 (48)
Asthenia (General disorders) | 34 (38)
Pyrexia (General disorders) | 24 (24)
Oedema (General disorders) | 22 (23)
Pain (General disorders) | 17 (17)
Malaise (General disorders) | 9 (9)
Chills (General disorders) | 6 (7)
Face oedema (General disorders) | 6 (6)
Disease progression (General disorders) | 5 (5)
Feeling hot (General disorders) | 4 (4)
Peripheral swelling (General disorders) | 4 (4)
Effusion (General disorders) | 3 (3)
Exercise tolerance decreased (General disorders) | 3 (3)
Feeling cold (General disorders) | 3 (3)
Multiple organ dysfunction syndrome (General disorders) | 3 (3)
Non-cardiac chest pain (General disorders) | 3 (3)
Calcinosis (General disorders) | 2 (2)
Generalised oedema (General disorders) | 2 (2)
Sudden death (General disorders) | 2 (2)
Swelling (General disorders) | 2 (2)
Swelling face (General disorders) | 2 (2)
Adverse drug reaction (General disorders) | 1 (1)
Axillary pain (General disorders) | 1 (1)
Early satiety (General disorders) | 1 (1)
Hypothermia (General disorders) | 1 (1)
Inflammation (General disorders) | 1 (1)
Influenza like illness (General disorders) | 1 (1)
Injection site pain (General disorders) | 1 (1)
Polyp (General disorders) | 1 (1)
Sudden cardiac death (General disorders) | 1 (1)
Ulcer (General disorders) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 14 (15)
Cholelithiasis (Hepatobiliary disorders) | 6 (6)
Cholecystitis acute (Hepatobiliary disorders) | 5 (5)
Hepatic cirrhosis (Hepatobiliary disorders) | 5 (5)
Hepatic steatosis (Hepatobiliary disorders) | 4 (4)
Cholecystitis chronic (Hepatobiliary disorders) | 3 (3)
Congestive hepatopathy (Hepatobiliary disorders) | 3 (3)
Hepatic failure (Hepatobiliary disorders) | 3 (3)
Hyperbilirubinaemia (Hepatobiliary disorders) | 3 (3)
Cholestasis (Hepatobiliary disorders) | 2 (2)
Hepatic cyst (Hepatobiliary disorders) | 2 (2)
Hepatic mass (Hepatobiliary disorders) | 2 (2)
Acute hepatic failure (Hepatobiliary disorders) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 1 (1)
Biliary tract disorder (Hepatobiliary disorders) | 1 (2)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Hepatic calcification (Hepatobiliary disorders) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 1 (1)
Hepatomegaly (Hepatobiliary disorders) | 1 (1)
Liver injury (Hepatobiliary disorders) | 1 (1)
Nonalcoholic fatty liver disease (Hepatobiliary disorders) | 1 (1)
Portal hypertension (Hepatobiliary disorders) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1)
Steatohepatitis (Hepatobiliary disorders) | 1 (1)
Subcapsular hepatic haematoma (Hepatobiliary disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 5 (6)
Seasonal allergy (Immune system disorders) | 5 (5)
Atopy (Immune system disorders) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (2)
Immune system disorder (Immune system disorders) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 116 (160)
Nasopharyngitis (Infections and infestations) | 61 (85)
Pneumonia (Infections and infestations) | 50 (59)
Bronchitis (Infections and infestations) | 31 (41)
Urinary tract infection (Infections and infestations) | 30 (37)
Gastroenteritis (Infections and infestations) | 20 (23)
Pharyngitis (Infections and infestations) | 19 (27)
Respiratory tract infection (Infections and infestations) | 17 (23)
Influenza (Infections and infestations) | 16 (18)
Sinusitis (Infections and infestations) | 14 (17)
COVID-19 (Infections and infestations) | 12 (12)
Cellulitis (Infections and infestations) | 9 (9)
Rhinitis (Infections and infestations) | 9 (9)
Septic shock (Infections and infestations) | 9 (9)
Lower respiratory tract infection (Infections and infestations) | 7 (7)
Vaginal infection (Infections and infestations) | 7 (7)
Herpes zoster (Infections and infestations) | 6 (6)
Gastrointestinal infection (Infections and infestations) | 5 (5)
Pharyngitis bacterial (Infections and infestations) | 5 (5)
Sepsis (Infections and infestations) | 5 (5)
Appendicitis (Infections and infestations) | 4 (6)
Cystitis (Infections and infestations) | 4 (4)
Gingivitis (Infections and infestations) | 4 (4)
COVID-19 pneumonia (Infections and infestations) | 3 (3)
Laryngitis (Infections and infestations) | 3 (3)
Tonsillitis (Infections and infestations) | 3 (3)
Clostridium difficile colitis (Infections and infestations) | 2 (2)
Clostridium difficile infection (Infections and infestations) | 2 (2)
Conjunctivitis (Infections and infestations) | 2 (2)
Helicobacter infection (Infections and infestations) | 2 (2)
Herpes simplex (Infections and infestations) | 2 (2)
Localised infection (Infections and infestations) | 2 (2)
Oral candidiasis (Infections and infestations) | 2 (2)
Otitis media (Infections and infestations) | 2 (3)
Pericoronitis (Infections and infestations) | 2 (2)
Peritonitis (Infections and infestations) | 2 (2)
Pharyngitis streptococcal (Infections and infestations) | 2 (2)
Tooth abscess (Infections and infestations) | 2 (2)
Urinary tract infection bacterial (Infections and infestations) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2)
Bacteraemia (Infections and infestations) | 1 (1)
Bacterial translocation (Infections and infestations) | 1 (1)
Bed bug infestation (Infections and infestations) | 1 (1)
Body tinea (Infections and infestations) | 1 (1)
Bronchiolitis (Infections and infestations) | 1 (1)
Campylobacter infection (Infections and infestations) | 1 (1)
Candida infection (Infections and infestations) | 1 (2)
Cat scratch disease (Infections and infestations) | 1 (1)
Cholecystitis infective (Infections and infestations) | 1 (1)
Chronic sinusitis (Infections and infestations) | 1 (1)
Conjunctivitis bacterial (Infections and infestations) | 1 (1)
Diarrhoea infectious (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (7)
Ear infection (Infections and infestations) | 1 (1)
Enteritis infectious (Infections and infestations) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1)
Eye infection (Infections and infestations) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1)
Gangrene (Infections and infestations) | 1 (1)
Gastroenteritis bacterial (Infections and infestations) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Hepatitis A (Infections and infestations) | 1 (1)
Hepatitis B (Infections and infestations) | 1 (1)
Hepatitis C (Infections and infestations) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1)
Impetigo (Infections and infestations) | 1 (1)
Infected cyst (Infections and infestations) | 1 (1)
Infected skin ulcer (Infections and infestations) | 1 (1)
Infective exacerbation of bronchiectasis (Infections and infestations) | 1 (1)
Lymphadenitis bacterial (Infections and infestations) | 1 (1)
Meningitis listeria (Infections and infestations) | 1 (1)
Metapneumovirus infection (Infections and infestations) | 1 (1)
Onychomycosis (Infections and infestations) | 1 (1)
Ophthalmic herpes zoster (Infections and infestations) | 1 (1)
Pelvic inflammatory disease (Infections and infestations) | 1 (1)
Periodontitis (Infections and infestations) | 1 (1)
Pharyngotonsillitis (Infections and infestations) | 1 (1)
Pneumonia influenzal (Infections and infestations) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1)
Pulpitis dental (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Sialoadenitis (Infections and infestations) | 1 (1)
Sinusitis bacterial (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (2)
Staphylococcal sepsis (Infections and infestations) | 1 (1)
Tonsillitis bacterial (Infections and infestations) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Urethritis (Infections and infestations) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1)
Viral pharyngitis (Infections and infestations) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 11 (11)
Contusion (Injury, poisoning and procedural complications) | 9 (10)
Fall (Injury, poisoning and procedural complications) | 5 (6)
Hand fracture (Injury, poisoning and procedural complications) | 4 (4)
Skin laceration (Injury, poisoning and procedural complications) | 4 (4)
Tooth fracture (Injury, poisoning and procedural complications) | 3 (3)
Animal bite (Injury, poisoning and procedural complications) | 2 (2)
Foot fracture (Injury, poisoning and procedural complications) | 2 (2)
Joint injury (Injury, poisoning and procedural complications) | 2 (2)
Skin injury (Injury, poisoning and procedural complications) | 2 (2)
Soft tissue injury (Injury, poisoning and procedural complications) | 2 (2)
Spinal fracture (Injury, poisoning and procedural complications) | 2 (2)
Upper limb fracture (Injury, poisoning and procedural complications) | 2 (2)
Wound (Injury, poisoning and procedural complications) | 2 (3)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1)
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Bone contusion (Injury, poisoning and procedural complications) | 1 (1)
Buttock injury (Injury, poisoning and procedural complications) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 1 (1)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Spinal column injury (Injury, poisoning and procedural complications) | 1 (1)
Splenic rupture (Injury, poisoning and procedural complications) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1)
Weight decreased (Investigations) | 25 (25)
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 15 (15)
Blood creatinine increased (Investigations) | 10 (10)
Platelet count decreased (Investigations) | 10 (10)
Weight increased (Investigations) | 9 (9)
Alanine aminotransferase increased (Investigations) | 8 (8)
Blood bilirubin increased (Investigations) | 8 (8)
Oxygen saturation decreased (Investigations) | 8 (8)
Aspartate aminotransferase increased (Investigations) | 7 (7)
Gamma-glutamyltransferase increased (Investigations) | 7 (7)
Haemoglobin decreased (Investigations) | 7 (7)
Blood potassium decreased (Investigations) | 6 (7)
Hepatic enzyme increased (Investigations) | 6 (6)
International normalised ratio increased (Investigations) | 5 (5)
Blood urea increased (Investigations) | 4 (4)
Brain natriuretic peptide increased (Investigations) | 4 (4)
Blood uric acid increased (Investigations) | 3 (3)
Electrocardiogram QT prolonged (Investigations) | 3 (3)
White blood cell count decreased (Investigations) | 3 (3)
Blood alkaline phosphatase increased (Investigations) | 2 (2)
Catheterisation cardiac (Investigations) | 2 (2)
Haemoglobin increased (Investigations) | 2 (2)
Heart rate increased (Investigations) | 2 (4)
Protein urine (Investigations) | 2 (2)
Protein urine present (Investigations) | 2 (2)
Vitamin D decreased (Investigations) | 2 (2)
Anticoagulation drug level above therapeutic (Investigations) | 1 (1)
Blood albumin increased (Investigations) | 1 (1)
Blood bicarbonate decreased (Investigations) | 1 (1)
Blood bilirubin unconjugated increased (Investigations) | 1 (1)
Blood immunoglobulin G increased (Investigations) | 1 (1)
Blood pressure decreased (Investigations) | 1 (1)
Blood pressure increased (Investigations) | 1 (1)
Blood thyroid stimulating hormone decreased (Investigations) | 1 (1)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1)
Blood triglycerides increased (Investigations) | 1 (1)
Blood urine (Investigations) | 1 (1)
C-reactive protein increased (Investigations) | 1 (1)
Cardiac output increased (Investigations) | 1 (1)
Coagulation time prolonged (Investigations) | 1 (1)
Ejection fraction decreased (Investigations) | 1 (1)
Electrocardiogram P wave abnormal (Investigations) | 1 (1)
Electrocardiogram ST-T change (Investigations) | 1 (1)
Electrocardiogram abnormal (Investigations) | 1 (1)
Fibrin D dimer increased (Investigations) | 1 (1)
Haematocrit decreased (Investigations) | 1 (1)
Heart rate decreased (Investigations) | 1 (1)
Heart sounds abnormal (Investigations) | 1 (1)
Liver function test abnormal (Investigations) | 1 (1)
Lymphocyte morphology abnormal (Investigations) | 1 (1)
Myocardial necrosis marker increased (Investigations) | 1 (1)
Occult blood (Investigations) | 1 (1)
Platelet count increased (Investigations) | 1 (1)
QRS axis abnormal (Investigations) | 1 (1)
Red blood cells urine (Investigations) | 1 (1)
Serum ferritin decreased (Investigations) | 1 (1)
Thyroxine free decreased (Investigations) | 1 (1)
Transaminases increased (Investigations) | 1 (2)
Troponin T increased (Investigations) | 1 (1)
Urine output decreased (Investigations) | 1 (1)
Vitamin B12 decreased (Investigations) | 1 (1)
White blood cell count increased (Investigations) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 50 (56)
Decreased appetite (Metabolism and nutrition disorders) | 41 (43)
Hyperuricaemia (Metabolism and nutrition disorders) | 17 (17)
Gout (Metabolism and nutrition disorders) | 15 (15)
Iron deficiency (Metabolism and nutrition disorders) | 12 (13)
Fluid retention (Metabolism and nutrition disorders) | 11 (12)
Hyponatraemia (Metabolism and nutrition disorders) | 7 (7)
Dehydration (Metabolism and nutrition disorders) | 5 (6)
Dyslipidaemia (Metabolism and nutrition disorders) | 5 (5)
Electrolyte imbalance (Metabolism and nutrition disorders) | 5 (6)
Fluid overload (Metabolism and nutrition disorders) | 4 (7)
Hyperlipidaemia (Metabolism and nutrition disorders) | 4 (4)
Diabetes mellitus (Metabolism and nutrition disorders) | 3 (3)
Folate deficiency (Metabolism and nutrition disorders) | 3 (4)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (3)
Overweight (Metabolism and nutrition disorders) | 3 (3)
Cachexia (Metabolism and nutrition disorders) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (3)
Hypoproteinaemia (Metabolism and nutrition disorders) | 2 (2)
Insulin resistance (Metabolism and nutrition disorders) | 2 (2)
Malnutrition (Metabolism and nutrition disorders) | 2 (2)
Metabolic acidosis (Metabolism and nutrition disorders) | 2 (2)
Obesity (Metabolism and nutrition disorders) | 2 (2)
Vitamin D deficiency (Metabolism and nutrition disorders) | 2 (2)
Calciphylaxis (Metabolism and nutrition disorders) | 1 (1)
Fructose intolerance (Metabolism and nutrition disorders) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1)
Lactose intolerance (Metabolism and nutrition disorders) | 1 (1)
Metabolic alkalosis (Metabolism and nutrition disorders) | 1 (1)
Steroid diabetes (Metabolism and nutrition disorders) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Vitamin B complex deficiency (Metabolism and nutrition disorders) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 103 (106)
Myalgia (Musculoskeletal and connective tissue disorders) | 78 (82)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 78 (90)
Arthralgia (Musculoskeletal and connective tissue disorders) | 57 (69)
Back pain (Musculoskeletal and connective tissue disorders) | 41 (45)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 (7)
Neck pain (Musculoskeletal and connective tissue disorders) | 7 (7)
Arthritis (Musculoskeletal and connective tissue disorders) | 5 (6)
Bone pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5 (5)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 (5)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 5 (6)
Tendonitis (Musculoskeletal and connective tissue disorders) | 5 (5)
Joint swelling (Musculoskeletal and connective tissue disorders) | 4 (4)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 4 (4)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 4 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 3 (3)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 3 (3)
Costochondritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2)
Mixed connective tissue disease (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 (2)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 2 (2)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Clubbing (Musculoskeletal and connective tissue disorders) | 1 (1)
Enthesopathy (Musculoskeletal and connective tissue disorders) | 1 (1)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Fracture malunion (Musculoskeletal and connective tissue disorders) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Myopathy (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 (1)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1)
Undifferentiated connective tissue disease (Musculoskeletal and connective tissue disorders) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3)
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bladder transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hepatic cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (4)
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neurofibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
POEMS syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Teratoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Headache (Nervous system disorders) | 328 (348)
Dizziness (Nervous system disorders) | 120 (131)
Syncope (Nervous system disorders) | 18 (19)
Hypoaesthesia (Nervous system disorders) | 14 (15)
Paraesthesia (Nervous system disorders) | 11 (12)
Presyncope (Nervous system disorders) | 11 (11)
Somnolence (Nervous system disorders) | 6 (6)
Head discomfort (Nervous system disorders) | 5 (5)
Memory impairment (Nervous system disorders) | 4 (4)
Restless legs syndrome (Nervous system disorders) | 4 (4)
Amnesia (Nervous system disorders) | 3 (3)
Migraine (Nervous system disorders) | 3 (4)
Cerebrovascular accident (Nervous system disorders) | 2 (2)
Neuralgia (Nervous system disorders) | 2 (2)
Neuropathy peripheral (Nervous system disorders) | 2 (2)
Sciatica (Nervous system disorders) | 2 (2)
Tremor (Nervous system disorders) | 2 (2)
Aphasia (Nervous system disorders) | 1 (1)
Brain injury (Nervous system disorders) | 1 (1)
Coma (Nervous system disorders) | 1 (1)
Disturbance in attention (Nervous system disorders) | 1 (1)
Dizziness exertional (Nervous system disorders) | 1 (1)
Dizziness postural (Nervous system disorders) | 1 (2)
Facial paralysis (Nervous system disorders) | 1 (1)
Hand-arm vibration syndrome (Nervous system disorders) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 1 (1)
Hyperaesthesia (Nervous system disorders) | 1 (1)
Intention tremor (Nervous system disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1)
Mental impairment (Nervous system disorders) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 1 (1)
Muscle contractions involuntary (Nervous system disorders) | 1 (1)
Nerve compression (Nervous system disorders) | 1 (1)
Post herpetic neuralgia (Nervous system disorders) | 1 (1)
Sedation (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Spinal cord compression (Nervous system disorders) | 1 (1)
Vocal cord paralysis (Nervous system disorders) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Insomnia (Psychiatric disorders) | 40 (41)
Depression (Psychiatric disorders) | 22 (22)
Anxiety (Psychiatric disorders) | 10 (10)
Poor quality sleep (Psychiatric disorders) | 8 (8)
Sleep disorder (Psychiatric disorders) | 4 (4)
Agitation (Psychiatric disorders) | 3 (3)
Confusional state (Psychiatric disorders) | 2 (2)
Restlessness (Psychiatric disorders) | 2 (2)
Alcoholism (Psychiatric disorders) | 1 (1)
Anxiety disorder (Psychiatric disorders) | 1 (1)
Bipolar II disorder (Psychiatric disorders) | 1 (1)
Borderline personality disorder (Psychiatric disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Emotional distress (Psychiatric disorders) | 1 (1)
Major depression (Psychiatric disorders) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1)
Neurosis (Psychiatric disorders) | 1 (1)
Panic attack (Psychiatric disorders) | 1 (1)
Stress (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 14 (16)
Proteinuria (Renal and urinary disorders) | 12 (12)
Renal failure (Renal and urinary disorders) | 10 (10)
Haematuria (Renal and urinary disorders) | 6 (7)
Chronic kidney disease (Renal and urinary disorders) | 5 (5)
Nephrolithiasis (Renal and urinary disorders) | 5 (5)
Dysuria (Renal and urinary disorders) | 3 (4)
Renal impairment (Renal and urinary disorders) | 3 (3)
Diabetic nephropathy (Renal and urinary disorders) | 2 (2)
Lupus nephritis (Renal and urinary disorders) | 2 (3)
Oliguria (Renal and urinary disorders) | 2 (2)
Pollakiuria (Renal and urinary disorders) | 2 (2)
Bladder spasm (Renal and urinary disorders) | 1 (1)
Focal segmental glomerulosclerosis (Renal and urinary disorders) | 1 (1)
Glomerulonephritis acute (Renal and urinary disorders) | 1 (2)
Hydronephrosis (Renal and urinary disorders) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 1 (1)
Nephropathy (Renal and urinary disorders) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1)
Renal cyst (Renal and urinary disorders) | 1 (1)
Renal pain (Renal and urinary disorders) | 1 (1)
Renal vasculitis (Renal and urinary disorders) | 1 (1)
Scleroderma renal crisis (Renal and urinary disorders) | 1 (1)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1)
Urinary bladder polyp (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 1 (1)
Urine abnormality (Renal and urinary disorders) | 1 (1)
Urine flow decreased (Renal and urinary disorders) | 1 (1)
Menstrual disorder (Reproductive system and breast disorders) | 8 (8)
Menstruation irregular (Reproductive system and breast disorders) | 6 (6)
Breast mass (Reproductive system and breast disorders) | 4 (5)
Ovarian cyst (Reproductive system and breast disorders) | 3 (3)
Pelvic fluid collection (Reproductive system and breast disorders) | 3 (3)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 (2)
Breast pain (Reproductive system and breast disorders) | 2 (2)
Fibrocystic breast disease (Reproductive system and breast disorders) | 2 (2)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 2 (2)
Adnexa uteri mass (Reproductive system and breast disorders) | 1 (1)
Amenorrhoea (Reproductive system and breast disorders) | 1 (1)
Breast calcifications (Reproductive system and breast disorders) | 1 (1)
Breast cyst (Reproductive system and breast disorders) | 1 (1)
Breast hyperplasia (Reproductive system and breast disorders) | 1 (1)
Breast swelling (Reproductive system and breast disorders) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1)
Gynaecomastia (Reproductive system and breast disorders) | 1 (1)
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 1 (1)
Hypomenorrhoea (Reproductive system and breast disorders) | 1 (1)
Intermenstrual bleeding (Reproductive system and breast disorders) | 1 (2)
Nipple pain (Reproductive system and breast disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Polycystic ovaries (Reproductive system and breast disorders) | 1 (1)
Prostatic calcification (Reproductive system and breast disorders) | 1 (1)
Prostatomegaly (Reproductive system and breast disorders) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 113 (131)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 103 (147)
Cough (Respiratory, thoracic and mediastinal disorders) | 72 (76)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 24 (26)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 19 (19)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 17 (17)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 17 (20)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 16 (17)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 15 (16)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 10 (10)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 9 (10)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Asthma (Respiratory, thoracic and mediastinal disorders) | 6 (10)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnoea paroxysmal nocturnal (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngeal cyst (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ventilation perfusion mismatch (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vocal cord dysfunction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 20 (20)
Pruritus (Skin and subcutaneous tissue disorders) | 13 (13)
Erythema (Skin and subcutaneous tissue disorders) | 12 (13)
Alopecia (Skin and subcutaneous tissue disorders) | 11 (11)
Urticaria (Skin and subcutaneous tissue disorders) | 5 (5)
Ecchymosis (Skin and subcutaneous tissue disorders) | 4 (4)
Eczema (Skin and subcutaneous tissue disorders) | 4 (5)
Skin lesion (Skin and subcutaneous tissue disorders) | 4 (4)
Acne (Skin and subcutaneous tissue disorders) | 3 (3)
Dermatitis (Skin and subcutaneous tissue disorders) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 (3)
Skin ulcer (Skin and subcutaneous tissue disorders) | 3 (3)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 2 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (2)
Night sweats (Skin and subcutaneous tissue disorders) | 2 (2)
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 (3)
Alopecia areata (Skin and subcutaneous tissue disorders) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 1 (1)
Chloasma (Skin and subcutaneous tissue disorders) | 1 (1)
Cold sweat (Skin and subcutaneous tissue disorders) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatomyositis (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatosis (Skin and subcutaneous tissue disorders) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1)
Intertrigo (Skin and subcutaneous tissue disorders) | 1 (1)
Lichen planus (Skin and subcutaneous tissue disorders) | 1 (1)
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 (1)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (1)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 (1)
Skin fissures (Skin and subcutaneous tissue disorders) | 1 (1)
Skin mass (Skin and subcutaneous tissue disorders) | 1 (1)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Cardiac assistance device user (Social circumstances) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 4 (4)
Abortion induced (Surgical and medical procedures) | 2 (2)
Abdominal hernia repair (Surgical and medical procedures) | 1 (1)
Dacryocystorhinostomy (Surgical and medical procedures) | 1 (1)
Endodontic procedure (Surgical and medical procedures) | 1 (1)
Hernia repair (Surgical and medical procedures) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 1 (1)
Oxygen therapy (Surgical and medical procedures) | 1 (1)
Flushing (Vascular disorders) | 201 (204)
Hypotension (Vascular disorders) | 36 (42)
Hypertension (Vascular disorders) | 12 (12)
Hyperaemia (Vascular disorders) | 8 (8)
Haematoma (Vascular disorders) | 7 (8)
Hot flush (Vascular disorders) | 6 (7)
Peripheral venous disease (Vascular disorders) | 5 (5)
Cyanosis (Vascular disorders) | 4 (4)
Shock (Vascular disorders) | 3 (3)
Raynaud's phenomenon (Vascular disorders) | 2 (2)
Varicose vein (Vascular disorders) | 2 (2)
Angiodysplasia (Vascular disorders) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1)
Claudication of jaw muscles (Vascular disorders) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1)
Pallor (Vascular disorders) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1)
Peripheral coldness (Vascular disorders) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1)
Thrombophlebitis superficial (Vascular disorders) | 1 (1)
Vena cava thrombosis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol (2018-07-13): https://cdn.clinicaltrials.gov/large-docs/37/NCT01560637/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-15): https://cdn.clinicaltrials.gov/large-docs/37/NCT01560637/SAP_001.pdf
  • Informed Consent Form (2018-07-13): https://cdn.clinicaltrials.gov/large-docs/37/NCT01560637/ICF_002.pdf